CLINICAL TRIAL: NCT03877640
Title: A Double-Blind, Sham Controlled Prospective Pilot Study of Urinary Stress Incontinence and Urgency in Women After 6 Treatments With HIFEM Technology (BTL EMSELLA)
Brief Title: Urinary Stress Incontinence and Urgency in Women With EMSELLA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Diego Sexual Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SDSM-2018-02
Record Dates: First submitted 2019-01-30; First posted 2019-03-18 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Stress Urinary Incontinence; Urge Incontinence
Keywords: incontinence; stress urgency incontinence; urge incontinence; EMSELLA
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence, Urge

STUDY DESIGN:
Intervention Model Description: Active and sham arms 2:1 run parallel. Upon completion, sham patients repeat visits with open label treatment.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Three blinded protocols available on the device, so care provider will not know to which treatment subject is randomized. Active treatment is not blinded for use in open label portion of study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active EMSELLA treatment (Active Comparator): 6 treatments on the BTL EMSELLA using a device protocol that is active HIFEM technology
  Interventions: Device: BTL EMSELLA
- Sham EMSELLA treatment (Sham Comparator): 6 treatments on the BTL EMSELLA with a sham device protocol that provides some sensation without active HIFEM technology
  Interventions: Device: BTL EMSELLA

INTERVENTIONS:
Device: BTL EMSELLA — High intensity focused electromagnetic (HIFEM) technology induces deep pelvic floor muscle contractions designed to deliver the equivalent of 11,200 Kegel exercises over 28 minutes.

SUMMARY:
The purpose of this prospective study is to examine the safety and efficacy of high intensity focused electromagnetic (HIFEM) technology for the treatment of women with stress urinary incontinence (SUI), urge incontinence (UI) and mixed stress urinary and urge incontinence (MUI), looking at any potential sexual health benefits that may be concomitantly achieved from this treatment.

DETAILED DESCRIPTION:
This is a blinded study to be conducted at San Diego Sexual Medicine in San Diego, CA. Participants meeting inclusion and exclusion criteria will receive one treatment cycle of active treatment or sham. The device will be equipped with 3 protocols in addition to the standard protocol, two of which are identical to the standard protocol (for active treatment) and one of which does not deliver HIFEM (for sham treatment). The active treatment arm consists of 6 treatments, 2 per week, with at least one day in between. Follow-up visits will occur at 4 weeks and 12 weeks after the last treatment. Unblinding will take place at the 12 week follow up visit, and subjects assigned to the sham arm will be crossed over to active treatment, beginning their first treatment on that day, completing 6 treatments and 2 follow up visits. Once unblinded the subject will be treated with the standard protocol of the device.

After the informed consent is signed, and inclusion and exclusion criteria completed, participants will complete validated questionnaires and undergo a baseline physical therapy assessment of pelvic floor muscle strength.

ELIGIBILITY:
Inclusion Criteria:

1. Subject provides written informed consent and HIPAA authorization before any study procedures are conducted;
2. Subject is female;
3. Subject is aged 21-80 years;
4. Subject has a body mass index (BMI) < 37 kg/m2;
5. Subject has stress urinary incontinence, urge incontinence, or mixed urinary incontinence as determined by the QUID;
6. Subject is currently sexually active and willing to continue sexual activity throughout the study;
7. Subject is willing to continue level of core exercise currently being performed or not performed during the study (e.g. gym, Pilates, yoga);
8. Subject is willing to maintain her current prescription and over the counter medications throughout the study without changing them;
9. Subject agrees to comply with the study procedures and visits.

Exclusion Criteria:

1. Subject has used the BTL EMSELLA device previously;
2. Subject has any significant pelvic organ prolapse;
3. Subject has clinically significant findings on physical examination;
4. Subject has any chronic medical condition (e.g. neurologic disorder) or psychologic disorder that the Principal Investigator feels makes her ineligible for the study;
5. Subject is unwilling to maintain current level of exercise throughout the study;
6. Subject has been diagnosed with overactive bladder or interstitial cystitis;
7. Subject experiences bladder pain or scores above 0 on the pain questions on the O'Leary/Sant Voiding and Pain Indices (ICSI/ICPI);
8. Subject experiences pain with sexual activity
9. Subject answers anything other than "almost never or never" or "a few times" on pain questions 17 or 18 of the Female Sexual Function Index (FSFI)
10. Subject answers anything other than "very low or none at all" or "low" on pain questions 19 of the (FSFI)
11. Subject planning to have surgery during the study;
12. Subject has untreated malignancy;
13. Subject is pregnant, planning to get pregnant or within 3 months postpartum;
14. Subject has a pacemaker;
15. Subject has and implant or IUD containing metal (e.g. copper 7);
16. Subject has piercing between the waist and knees and is not willing to remove it before each treatment;
17. Subject has a history of substance abuse within 12 months prior, or consuming > 14 alcoholic drinks per week;
18. Subject has received an investigational drug within 30 days prior to signing consent;
19. Subject has any condition or exhibits behavior that indicates to the Principal Investigator that the Subject is unlikely to be compliant with study procedures and visits.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — cis-gender woman
Enrollment: 21 (Estimated)
Dates: Start 2019-01-11 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to 18 weeks for active arm; up to 32 weeks for sham arm
  Serious adverse events and adverse events related to device will be collected to assess safety
QUID (Questionnaire for Urinary Incontinence Diagnosis) | At screen, 4 weeks, 6 weeks, 10 weeks, 18 weeks; for sham arm additionally at 20 weeks, 24 weeks, 32 weeks
  Change in Questionnaire for Urinary Incontinence Diagnosis (QUID) from pre-treatment to each follow up visit

SECONDARY OUTCOMES:
FSFI (Female Sexual Function Index) Orgasm Domain | At screen, 4 weeks, 6 weeks, 10 weeks, 18 weeks; for sham arm additionally at 20 weeks, 24 weeks, 32 weeks
  Change in Orgasm Domain of the Female Sexual Function Index from pre-treatment to follow up visits. Range is 0-6 with higher the results representing better outcome
FSFI (Female Sexual Function Index) | At screen, 4 weeks, 6 weeks, 10 weeks, 18 weeks; for sham arm additionally at 20 weeks, 24 weeks, 32 weeks
  Change in total score of the Female Sexual Function Index from pre-treatment to follow up visits. Range is 2-36, with higher results representing better the outcome, and 26.55 and above signifying no sexual dysfunction
FSDS-DAO (Female Sexual Distress Score-Desire, Arousal, Orgasm) | At screen, 4 weeks, 6 weeks, 10 weeks, 18 weeks; for sham arm additionally at 20 weeks, 24 weeks, 32 weeks
  Change in total score of the Female Sexual Distress Score-Desire, Arousal, Orgasm from pre-treatment to follow up visits. Range is from 0-60 with lower results representing the better outcome.
ISCI (Interstitial Cystitis Symptoms Index )/ICPI (Interstitial Cystitis Problem Index) | At screen, 4 weeks, 6 weeks, 10 weeks, 18 weeks; for sham arm additionally at 20 weeks, 24 weeks, 32 weeks
  Change in total score of the ICSI/ICPI Questionnaire from pre-treatment to follow up visits. Range is 0-35, with lower results representing the better the outcome.
Modified Oxford Scale measuring pelvic floor strength | At screen, 10 weeks, 18 weeks; for sham arm additionally at 24 weeks, 32 weeks
  Change in degree of force based on the modified Oxford scale measuring pelvic floor muscle strength from pre-treatment to follow up visits. Scale is a single recording from 0 (lack of muscle response) to 5 (strong contraction, firm compression) with higher results representing the better the outcome.

OTHER OUTCOMES:
PGI-I (Patient global impression of improvement) | At 18 weeks; for sham arm additionally at 32 weeks
  Patient global impression of improvement, range 2-14, with higher results representing the better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sue W Goldstein, BA, Study Director — Clinical Research Manager
Locations (1):
- San Diego Sexual Medicine, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almeida FG, Bruschini H, Srougi M. Urodynamic and clinical evaluation of 91 female patients with urinary incontinence treated with perineal magnetic stimulation: 1-year followup. J Urol. 2004 Apr;171(4):1571-4; discussion 1574-5. doi: 10.1097/01.ju.0000117791.72151.f8. PMID 15017223
- [Background] Coletti D, Teodori L, Albertini MC, Rocchi M, Pristera A, Fini M, Molinaro M, Adamo S. Static magnetic fields enhance skeletal muscle differentiation in vitro by improving myoblast alignment. Cytometry A. 2007 Oct;71(10):846-56. doi: 10.1002/cyto.a.20447. PMID 17694560
- [Background] Ishikawa N, Suda S, Sasaki T, Yamanishi T, Hosaka H, Yasuda K, Ito H. Development of a non-invasive treatment system for urinary incontinence using a functional continuous magnetic stimulator (FCMS). Med Biol Eng Comput. 1998 Nov;36(6):704-10. doi: 10.1007/BF02518872. PMID 10367460
- [Background] Ostrovidov S, Hosseini V, Ahadian S, Fujie T, Parthiban SP, Ramalingam M, Bae H, Kaji H, Khademhosseini A. Skeletal muscle tissue engineering: methods to form skeletal myotubes and their applications. Tissue Eng Part B Rev. 2014 Oct;20(5):403-36. doi: 10.1089/ten.TEB.2013.0534. Epub 2014 Feb 24. PMID 24320971
- [Background] Stolting MN, Arnold AS, Haralampieva D, Handschin C, Sulser T, Eberli D. Magnetic stimulation supports muscle and nerve regeneration after trauma in mice. Muscle Nerve. 2016 Apr;53(4):598-607. doi: 10.1002/mus.24780. PMID 26202157
- [Background] Truijen G, Wyndaele JJ, Weyler J. Conservative treatment of stress urinary incontinence in women: who will benefit? Int Urogynecol J Pelvic Floor Dysfunct. 2001;12(6):386-90. doi: 10.1007/s001920170018. PMID 11795642
- [Background] Wallis MC, Davies EA, Thalib L, Griffiths S. Pelvic static magnetic stimulation to control urinary incontinence in older women: a randomized controlled trial. Clin Med Res. 2012 Feb;10(1):7-14. doi: 10.3121/cmr.2011.1008. Epub 2011 Aug 4. PMID 21817123
- [Background] Yamanishi T, Yasuda K, Suda S, Ishikawa N, Sakakibara R, Hattori T. Effect of functional continuous magnetic stimulation for urinary incontinence. J Urol. 2000 Feb;163(2):456-9. PMID 10647653
- [Background] Yamanishi T, Yasuda K, Sakakibara R, Hattori T, Ito H, Murakami S. Pelvic floor electrical stimulation in the treatment of stress incontinence: an investigational study and a placebo controlled double-blind trial. J Urol. 1997 Dec;158(6):2127-31. doi: 10.1016/s0022-5347(01)68176-x. PMID 9366328
- [Background] Yang SS, Jee S, Hwang SL, Sohn MK. Strengthening of Quadriceps by Neuromuscular Magnetic Stimulation in Healthy Subjects. PM R. 2017 Aug;9(8):767-773. doi: 10.1016/j.pmrj.2016.12.002. Epub 2017 Jan 8. PMID 28082179

DOCUMENTS (1):
  • Informed Consent Form (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT03877640/ICF_000.pdf